CLINICAL TRIAL: NCT03575052
Title: A Phase 3b, Multicenter, Randomized, Double-blind, Placebo-controlled, Safety Study of Pimavanserin Therapy in Adult and Elderly Subjects Experiencing Neuropsychiatric Symptoms Related to Neurodegenerative Disease
Brief Title: A Safety Study of Pimavanserin in Adult and Elderly Subjects Experiencing Neuropsychiatric Symptoms Related to Neurodegenerative Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-046; 2017-003536-36 (EudraCT Number)
Record Dates: First submitted 2018-06-09; First posted 2018-07-02 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Neuropsychiatric Symptoms Related to Neurodegenerative Disease
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug - Pimavanserin (Experimental)
  Interventions: Drug: Pimavanserin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg total daily dose, tablets, once daily by mouth (provided as two 17 mg NUPLAZID® tablets)
  Arms: Drug - Pimavanserin
Drug: Placebo — Placebo, tablets, once daily by mouth (provided as two placebo tablets)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of pimavanserin compared to placebo in adult and elderly subjects with neuropsychiatric symptoms related to neurodegenerative disease.

ELIGIBILITY:
Inclusion Criteria:

1. Can understand the nature of the trial and protocol requirements and provide written informed consent. If the subject is deemed not competent to provide informed consent, the following requirements for consent must be met:

   1. The subject's legally acceptable representative (LAR) (or study partner/caregiver, if local regulations allow) must provide written informed consent
   2. The subject must provide written (if capable) informed assent
2. Subject requires some or complete assistance with one or more of the following:

   1. Instrumental activities of daily living (communication, transportation, meal preparation, shopping, housework, managing medications, managing personal finances) OR
   2. Basic activities of daily living (personal hygiene, dressing, eating, maintaining continence or transferring)
3. Meets clinical criteria for at least one of the following disorders, with or without cerebrovascular disease (CVD):

   1. Parkinson's disease with or without dementia as defined by the Movement Disorder Society's Task Force
   2. Dementia with Lewy bodies (DLB)
   3. All-cause dementia, possible or probable Alzheimer's disease (AD)
   4. Frontotemporal degeneration spectrum disorders, including possible or probable:

   i. Behavioral variant frontotemporal dementia

   ii. Progressive supranuclear palsy

   iii. Corticobasal degeneration

   e. Vascular dementia, including post-stroke dementia multi-infarct dementia and/or subcortical ischemic vascular dementia (SIVD)
4. Has a designated study partner/caregiver
5. Can come to the clinic for study visits with a study partner/caregiver
6. If the subject is female, she must not be pregnant or breastfeeding. She must also be of non-childbearing potential (defined as either surgically sterilized or at least 1 year postmenopausal) or must agree to use a clinically acceptable method of contraception or be abstinent.
7. If the subject is taking an antipsychotic medication at the time of screening, the antipsychotic medication must be discontinued 2 weeks or 5 half-lives (whichever is longer)

Exclusion Criteria:

1. Is in hospice, is receiving end-of-life palliative care, or is bedridden
2. Has psychotic symptoms that are primarily attributable to delirium or substance abuse (i.e., neuropsychiatric symptoms not related to neurodegenerative disease)
3. Has current evidence of an unstable neurological, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies that, in the judgment of the Investigator, would jeopardize the safe participation of the subject in the study or significantly interfere with the conduct or interpretation of the study
4. Has a known personal or family history of long QT syndrome or family history of sudden cardiac death
5. Has a clinical significant CNS abnormality that is most likely contributing to the dementia or findings on MRI or CT including:

   1. intracranial mass lesion
   2. vascular malformation
   3. evidence of >4 hemosiderin deposits
6. The urine drug screen result at Visit 1 (Screening) indicates the presence of amphetamine/methamphetamine, barbiturates, cocaine, or phencyclidine (PCP). Subjects who test positive for amphetamines and who have a valid prescription may be retested if they agree to abstain from the medication for the length of their participation in the study. The presence of benzodiazepines, marijuana (THC), or opiates does not necessarily exclude the subject from the study, as assessed by the Investigator in consultation with the Medical Monitor.
7. Has previously been enrolled in any prior clinical study with pimavanserin or is currently taking pimavanserinIs judged by the Investigator or the Medical Monitor to be inappropriate for the study for any reason

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (104):
- United States (21):
  - Cognitive Clinical Trials, Gilbert, Arizona
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Syrentis Clinical Research, Santa Ana, California
  - Indago Research & Health Center Inc, Hialeah, Florida
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Global Medical Institutes, Miami, Florida
  - Future Care Solution, LLC, Miami, Florida
  - MediClear Medical & Research Center, Inc., Miami, Florida
  - Novel Clinical Research LLC, Miami, Florida
  - Laszlo J Mate, MD, PA, North Palm Beach, Florida
  - University of South Florida, Tampa, Florida
  - Synexus Clinical Research US, The Villages, Florida
  - Boston Center Memory, Newton, Massachusetts
  - Cognitive Clinical Trials LLC, Papillion, Nebraska
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - UNC Hospital, Chapel Hill, North Carolina
  - Insight Clinical Trials LLC, Shaker Heights, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Central for Biomedical Research, LLC, Knoxville, Tennessee
- Bulgaria (6):
  - Centre for Mental Health Prof. Dr. Ivan Temkov, Lazur Compl., Park Ezero, Burgas
  - UMHAT Psych clin for gen psychiatry and addictions, Pleven
  - DCC Sv. Vrach and Sv. Sv. Kozma and Damyan, Sofia
  - Diagnostic Consultative Centre, 2, N. Vaptzarov Street, Varna
  - Diagnostic Consultative Centre-Mladost-Psychiatry, 15, Republika Blvd, Varna
  - Mental Health Center Vratza EOOD, 1 Belasitsa St, Vratsa
- Colombia (4):
  - E.S.E. Hospital Mental de Antioquia, Bello, Antioquia
  - Centr Investigaciones y Proyectos en Neurociencias, Barranquilla, Atlántico
  - Psynapsis Salud Mental S.A., Pereira, Risaralda Department
  - Centro de Investigaciones del Sistema Nervioso, Bogotá
- Czechia (7):
  - BRAIN-SOULTHERAPY s.r.o., , Lekarna Jalta, Namesti Jana Masaryka 3113, Kladno
  - Fakultni nemocnice Olomouc, Olomouc
  - A-shine s.r.o./ Lekarna Centrum, Pilsen
  - AD71, s.r.o.,/Hostivarska Iekarna, Prague
  - Axon Clinical, Prague
  - Neuropsychiatrie, s.r.o., Lekarna 6ka, Fajtlova 1, Prague
  - AD71, s.r.o., /,Lekarna DPS Recruiting, Říčany
- Georgia (5):
  - Petre Sarajishvili Institute of Neurology LLC, Tbilisi
  - Pineo Medical Ecosystem LTD, Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
  - Health Institute LLC, Tbilisi
  - S. Khechinashvili University Hospital LLC, Tbilisi
- Mexico (5):
  - Hospital Universitario Saltillo, Saltillo, Coahuila
  - Instituto Nacional de Neurologia y Neurocirugia, Mexico City, Delegacion Tlalpan
  - Centro Regional para Adulto Mayor, Hsp Univ, JEG, Monterrey, Nuevo León
  - Clinicos y Especialidades Medicas, Monterrey, Nuevo León
  - Christus Muguerza Hospital Sur, Monterrey, Nuevo León
- Poland (13):
  - Neurologi ZOZ Cntr Leczenia SM Badan Klinicznych, Plewiska, Poznan
  - MlynowaMed SP Psych Dr. Joanna Lazarcyck, Bialystok
  - Wlokiennicza Me Sp Prak Lekarska Dromasz Markowski, Bialystok
  - Przychodnia Srodmiescie Sp. z.o.o., Bydgoszcz
  - ISPL Wieslaw Jerzy Cubala, Gdansk
  - NZOZ Wielospecjalistyczna Poradnia Lekarska Synap, Katowice
  - Silmedic Sp. z.o.o., Katowice
  - Krakowska Ak Neuro Sp.- Centrum Neuro Klinicznej, ul. Arianska 7/3, Krakow
  - Centrum Medyczne HCP Sp. z.o.o., Poznan
  - NZOZ Syntonia Poradnia Zdrowia Psychicznego, ul. Cyprysowa 2F/ 9,10, Pruszcz, Pruszcz Gdański
  - Neuro-Care Sp. z.o.o. sp. Komandytowa, Siemianowice Śląskie
  - Neuro-care, Siemianowice Śląskie
  - RCMed Oddzial Sochaczew, ul. _eromskiego 41A, Sochaczew
- Romania (4):
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca, Cluj
  - Spitalul clinic CF Constanta, Sectia Neurologie, Constanța
  - Med Anima SRL, Clinica de psihiatrie, Iași
  - S.C. Carpe Diem SRL, Sibiu
- Russia (13):
  - Regional Specialized Psychiatric Hospital #2, Tonnel’nyy, Kochubeev District
  - Federal Siberian Sci Clinical Center of Med and Bio, Krasnoyarsk, Krasnoyarksk Region
  - Clinic "Hundred Years", Tomsk, Tomsk Oblast
  - Mental Health Research Center, Moscow
  - City Clinical Hospital #34, Novosibirsk
  - Leningrad Regional Psychoneurological Dispensary, Roshchino
  - St. Nicholas the Wonder Worker Psychiatric Hospital, Saint Petersburg
  - FSBI NMRC PN n.a. V.M. Bekhterev, Saint Petersburg
  - City Psychiatric Hospital #3, Saint Petersburg
  - Samara Psychiatric Hospital, Samara
  - Saratov City Clinical Hospital V. I. Razumovsky, Saratov
  - Smolensk State Medical University, Smolensk
  - Stavropol Regional Clin Spec Psych Hospital #1, Stavropol
- Serbia (10):
  - CHC Dr Dragisa Misovic- Dedinje, Belgrade
  - Clinical Center of Serbia, Clinic for Psychiatry, Belgrade
  - Military Medical Academy, Belgrade
  - Clinic for Psychiatric Diseases Dr. Laza Lazarevic, Belgrade
  - Klinicki Centar Srbije (KCS)- Klinika za nerurologiju, Belgrade
  - Special Hospital for Psychiatric Diseases "Kovin", Kovin
  - Clinical Center Kragujevac, Clinic for Neurology, Kragujevac
  - Clinical Center Kragujevac, Clinic of Psychiatry, Kragujevac
  - Clinical Center Nis, Clinic for Psychiatry, Toponica
  - General Hospital Valjevo, Department for Neurology, Valjevo
- South Africa (3):
  - Neurology Practice, Pretoria, Gauteng
  - Dr. Stanley Lipshitz Clinic Inc., Sandton, Gauteng
  - Flexivest Fourteen Research Centre Potocnik F C V, Durbanville, Western Cape
- Ukraine (13):
  - Dnipr Regional Clinical Hospital n.a. Mechnikov, Dnipro
  - I.I. Mechnykov Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Dnipropetrovsk Regional Rehabilitation Hospital, Dnipro
  - Ivano-Frankivsk Nat Med Uni Dep Psychiatry, Regional Hospital, Ivano-Frankivsk
  - Institute of Neruology, Nat Acad of Med Sci of UKR, Kharkiv
  - Institute of Neurology, Kharkiv
  - Municipal Non-Commercial Institution of Kharkiv Regional Council "Kharkiv Regional Clinical Psychiatric Hospital # 3" 46, Ac. Pavlova str, Kharkiv
  - Kyiv Regional Medical Incorp. Psychiatria, Center, Kyiv
  - Kyiv Regional Psychiatric and Narcological Medical Association 8, Vokzalna str, Kyiv
  - Ternopil Regional Communal Clinical Psychoneurological Hospital 14, Troleibusna str., Ternopil
  - Municipal Institution "Vinnytsya Regional Psychoneurological Hospital n.a. Acad. O.I.Yushchenko", Male Department #7, Female Department #10, Vinnytsya, National Medical University n.a. M.I.Pyrogov, 109 Pyrogova str., Vinnytsia
  - Municipal Unst Zaporizhzhya Reg Clinical Hosp Neurology, Zaporizhzhya
  - Zaporizhzhya Reg. Hospital, Neurology Dpt, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alva G, Cubala WJ, Berrio A, Coate B, Abler V, Pathak S. Safety Profile of Pimavanserin Therapy in Elderly Patients with Neurodegenerative Disease-Related Neuropsychiatric Symptoms: A Phase 3B Study. J Alzheimers Dis. 2024;98(1):265-274. doi: 10.3233/JAD-231167. PMID 38427485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study in adult and elderly patients with neuropsychiatric symptoms related to neurodegenerative disease.
Groups:
- Placebo: Pimavanserin matching placebo (administered as 2 capsules) once daily
- Pimavanserin 34 mg: Pimavanserin 34 mg (administered as 2 x 17 mg capsules) once daily
Period: Overall Study
Arm/Group | Placebo | Pimavanserin 34 mg
Started | 392 | 392
Completed | 367 | 363
Not Completed | 25 | 29
Not completed — Adverse Event | 6 | 10
Not completed — Not further specified | 5 | 7
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 3 | 0
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Study drug noncompliance | 1 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomised
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pimavanserin 34 mg | Total
Number analyzed (Participants) | 392 | 392 | 784
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (7.13) | 72.7 (6.91) | 72.4 (7.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 240 | 453
  Male | 179 | 152 | 331
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 00 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 367 | 368 | 735
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  Colombia | 13 | 11 | 24
  Romania | 3 | 3 | 6
  United States | 117 | 115 | 232
  Czechia | 21 | 17 | 38
  Ukraine | 62 | 45 | 107
  Poland | 54 | 55 | 109
  Mexico | 6 | 8 | 14
  South Africa | 6 | 8 | 14
  Georgia | 8 | 19 | 27
  Russia | 55 | 55 | 110
  Bulgaria | 29 | 29 | 58
  Serbia | 18 | 27 | 45

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: Number (%) of patients with treatment-emergent AEs
Time Frame: Treatment Period: 8 weeks
Population: All patients randomised and treated
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pimavanserin 34 mg
Number analyzed (Participants) | 392 | 392
Participants | 115 | 119

2. Secondary Outcome: Change From Baseline to Week 8 in Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A)
Description: The ESRS is a questionnaire to assess drug induced movement disorders, including parkinsonism; the ESRS-A is an accepted modified form of the original ESRS. The ESRS-A consists of 4 subscales and 4 clinical global impression movement severity scales of Parkinsonism, dyskinesia, dystonia, and akathisia. The Parkinsonism scale consists of 10 items, the dyskinesia subscale of 6 items, the dystonia subscale of 6 items, and the akathisia subscale of 2 items. Each item is scored on a 6-point scale from 0 (absent) to 5 (extreme). The ESRS-A total score is the sum of the 24 item scores with a possible range of 0 to 120. Higher scores denote more severe drug-induced movement disorders.
Time Frame: Treatment Period: 8 weeks
Population: All patients randomised and treated
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pimavanserin 34 mg
Number analyzed (Participants) | 392 | 392
score on a scale | -0.6 (0.19) | -0.5 (0.19)

3. Secondary Outcome: Change From Baseline to Week 8 in Mini-Mental State Examination (MMSE)
Description: The MMSE is a 30-item questionnaire to quantitatively assess cognition, focusing on questions related to time and place of testing, repeating lists of words, arithmetic, language use and comprehension, and copying a drawing. Each of the 30 items has 2 possible values of 0 (incorrect) or 1 (correct). The MMSE total score is derived as the sum of the 30 item scores; thus, it can range from 0 to 30. Lower scores indicate more severe cognitive impairment.
Time Frame: Treatment Period: 8 weeks
Population: All patients randomised and treated
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pimavanserin 34 mg
Number analyzed (Participants) | 392 | 392
score on a scale | 1.2 (0.15) | 1.3 (0.15)

ADVERSE EVENTS:
Time Frame: Treatment period (8 weeks) and follow-up period (30 days): total of approximately 15 weeks
Arm/Group | Placebo | Pimavanserin 34 mg
All-Cause Mortality (participants affected / at risk) | 2/392 | 2/392
Serious Adverse Events (participants affected / at risk) | 6/392 | 8/392
Other Adverse Events (participants affected / at risk) | 16/392 | 25/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=392) | Pimavanserin 34 mg (N=392)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femure fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=392) | Pimavanserin 34 mg (N=392)
Urinary tract infection (Infections and infestations) | 16 (16) | 25 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03575052/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03575052/SAP_001.pdf